CLINICAL TRIAL: NCT04740346
Title: A Prospective Multi-center Randomized Clinical Trial to Compare Survival Rates and Quality of Life According to Follow-up Period in Patients Who Underwent Radical Gastrectomy for Advanced Gastric Cancer (STOFOLUP Trial)
Brief Title: Survival Rates and Quality of Life According to Follow-up Period After Gastrectomy for Gastric Cancer (STOFOLUP)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Collaborators: Korea Health Industry Development Institute (Other Government)
Responsible Party: Principal Investigator, Keun Won Ryu, Principal Investigator, National Cancer Center, Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HC20C0155
Record Dates: First submitted 2021-02-01; First posted 2021-02-05 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Gastric Cancer; Recurrence; Quality of Life
MeSH Terms: conditions — Stomach Neoplasms; Recurrence | interventions — Tomography, X-Ray Computed; Diagnostic Imaging; Hematologic Tests

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3 months follow-up (Experimental): Patients will be follow-up every 3 months after gastrectomy.
  Interventions: Diagnostic Test: Computed tomography, Chest X-ray, and blood test
- 6 months follow-up (Active Comparator): Patients will be follow-up every 6 months after gastrectomy.
  Interventions: Diagnostic Test: Computed tomography, Chest X-ray, and blood test

INTERVENTIONS:
Diagnostic Test: Computed tomography, Chest X-ray, and blood test — CT will be performed every 3 months after gastrectomy in the 3-months follow-up group. CT will be performed every 6 months after gastrectomy in the 6 months follow-up group.

SUMMARY:
This study is a multi-center, prospective, randomized controlled study. The aim of this study is to compare survival rates and to observe quality of life and nutritional status according to follow-up period in patients who underwent radical gastrectomy for stage 2 or 3 gastric cancer.

DETAILED DESCRIPTION:
The hypothesis of this study is that the survival rates would be different between the 3 months and 6 months follow-up groups. The investigators expected survival differences of 6% and the anticipated 3-year overall survival is 83% in the 6 months follow-up group based on the previous 3 phase clinical trial. On the basis of this hypothesis, the sample size was calculated as 886 patients.

Patients who were diagnosed as stage 2 or 3 gastric cancer after gastrectomy will be assigned to 3 months or 6 months follow-up group. The planned examinations including blood test, X-ray , CT, endoscopy, and nutritional markers will be performed according to the protocol and each patients will be followed up for 3 years after enrollment.

The primary endpoint is 3 year overall survival and secondary endpoints are other survivals such as 3-year disease-free survival and gastric cancer specific survival, quality of life, and nutritional parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 19 years or more
* Patients who are diagnosed with pathological stage II or III gastric adenocarcinoma according to the AJCC 8th edition
* Patients who can understand all information about the trial and decide for themselves whether to participate in this study

Exclusion Criteria:

* Vulnerable patients such as pregnant and intellectual disability
* Patients who cannot undergo CT owing to poor kidney function or severe adverse effects
* Patients who are already in another study and cannot follow the schedule for this trial
* Patients who are diagnosed with a cancer other than gastric cancer within five years before the gastrectomy
* Patients being treated for a cancer other than gastric cancer

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 886 (Estimated)
Dates: Start 2021-07-05 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
3-year overall survival | 3 years after surgery
  Death from any cause is defined as an event.

SECONDARY OUTCOMES:
3-year recurrence-free survival rate | 3 years after surgery
  Death from any cause and gastric cancer recurrence are an event.
3-year gastric cancer specific survival rate | 3 years after surgery
  Death from gastric cancer is the only event.
3-year post-recurrence survival rate | 3 years after surgery
  from recurrence detection date to last follow-up date (or death)
Summary score of KOQUSS-40 questionnaire | 3 years after surgery
  KOQUSS-40 consists of 8 domains with 40 questions for quality of life and post-gastrectomy symptoms. We will calculate the KOQUSS-40 summary score of each group and compare them between the two groups. The summary score is defined as the mean of eight symptom domains (Indigestion, dysphagia, reflux, dumping syndrome, bowel habit change, constipation, psychological factors, and worry about cancer). The minimum and maximum values are 0 and 100, and higher scores mean a better quality of life.
Summary score of EORTC QLQ C30 | 3 years after surgery
  EORTC QLQ C30 consists of 15 domains with 30 questions for quality of life of cancer patients. The 15 domains consist of five functional scales (physical, role, cognitive, emotional, and social functioning), a global QOL scale, three symptom scales (fatigue, nausea and vomiting, and pain), and six single items (appetite loss, diarrhea, dyspnea, constipation, insomnia, financial impact).
  We will calculate the EORTC QLQ C30 summary score of each group and compare them between the two groups. The summary score is defined as the mean of 13 domains (excluding global QOL scale and financial impact). The minimum and maximum values are 0 and 100, and higher scores mean a better quality of life.
Summary score of EORTC QLQ STO22 | 3 years after surgery
  EORTC QLQ STO22 consists of 9 domains with 22 questions for stomach cancer patients' symptoms. The 9 domains consist of five symptom scales (dysphagia, pain, reflux symptom, eating restriction, anxiety), four single items (having a dry mouth, taste, body image, and hair loss).
  We will calculate the EORTC QLQ STO22 summary score of each group and compare them between the two groups. The summary score is defined as the mean of 9 domains. The minimum and maximum values are 0 and 100, and higher scores mean a better quality of life.
Difference of body weight (kg) | 3 years after surgery
  Difference of body weight between preoperative and postoperative 3 year values
Incidence of iron deficiency anemia | 3 years after surgery
  Incidence of iron deficiency anemia for the 3 year follow-up after gastrectomy
Incidence of vitamin B12 deficiency | 3 years after surgery
  Incidence of vitamin B12 deficiency for the 3 year follow-up after gastrectomy

CONTACTS AND LOCATIONS:
Overall Officials: Keun Won Ryu, MD PhD, Principal Investigator — National Cancer Center, Korea
Locations (16):
- South Korea (16):
  - National Cancer Center, Korea, Goyang-si, Gyeonggi-do
  - Dongnam Institute of Radiological and Medical Sciences, Busan
  - Kosin University Gospel Hospital, Busan
  - Gyeongsang National University Changwon Hospital, Changwon
  - Keimyung University Dongsan Hospital, Daegu
  - Kyungpook National University Chilgok Hospital, Daegu
  - Chonnam National University Hwasun Hospital, Hwasun
  - Gyeongsang National University Hospital, Jinju
  - CHA Bundang Medical Center, Seongnam
  - Asan Medical Center, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Seoul St. Mary's Hospital, Seoul
  - Yonsei Univeristy College of Medicine, Seoul
  - Ajou University School of Medicine, Suwon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Eom BW, Koo DH, An JY, Lee HH, Kim HI, Hur H, Yoo MW, Ryu MH, Lee HJ, Kim SM, Park JH, Min JS, Seo KW, Jeong SH, Jeong O, Kwon OK, Ryu SW, Yoo CH, Bae JM, Ryu KW. Prospective multicentre randomised clinical trial comparing survival rates, quality of life and nutritional status between advanced gastric cancer patients with different follow-up intensities: study protocol for the STOFOLUP trial. BMJ Open. 2021 Dec 8;11(12):e056187. doi: 10.1136/bmjopen-2021-056187. PMID 34880028